CLINICAL TRIAL: NCT05408234
Title: Modified Foot Exercise to Improve Peripheral Perfussion and Sensitivity on Type 2 Diabetes Patients
Brief Title: Modified Foot Exercise to Improve Sensitivity and Perfussion on Type 2 Diabetes Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitas Sebelas Maret (Other)
Responsible Party: Principal Investigator, Nurhasan Agung Prabowo, Doctor, Universitas Sebelas Maret
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FootExercise
Record Dates: First submitted 2022-06-01; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: foot exercise, Diabetes Mellitus type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The study was conducted in the control and treatment groups where the control group will get the treatment of doing modified leg exercises for one week. The control group did not get the modified leg exercise. Both groups received standard therapy for type 2 diabetes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smart Foot Exercise (Experimental): The patient lies supine (supine) with the legs raised 450 while supported for 1-3 minutes until blanching occurs (the skin becomes pale).
  The patient sits on the edge of the bed with the legs hanging down and then performs dorsiflexion, plantarflexion, inversion, and eversion for 3 minutes until the skin appears red.
  The patient lies supine with the legs covered with a blanket for 3-5 minutes. This whole cycle is repeated 3-6 times per session, and each session is repeated 2-4 times a day.
  Movement using newspaper media, namely by:
  Place a sheet of newspaper on the floor, then shape the sheet into a ball with both feet.
  The ball shape is then opened into a sheet as before with both feet. Tear the newspaper into two parts, and separate the two parts of the newspaper. Tear the first newspaper into small pieces with both feet. Remove the bunch of stubs and place them in a second, whole newspaper. Wrap everything into a ball shape with both feet. This step is enough to do once.
  Interventions: Other: Smart Foot Exercise

INTERVENTIONS:
Other: Smart Foot Exercise — The patient lies supine (supine) with the legs raised 450 while supported for 1-3 minutes until blanching occurs (the skin becomes pale).
  The patient sits on the edge of the bed with the legs hanging down and then performs dorsiflexion, plantarflexion, inversion, and eversion for 3 minutes until the skin appears red.
  The patient lies supine with the legs covered with a blanket for 3-5 minutes. This whole cycle is repeated 3-6 times per session, and each session is repeated 2-4 times a day.
  Movement using newspaper media, namely by:
  Place a sheet of newspaper on the floor, then shape the sheet into a ball with both feet.
  The ball shape is then opened into a sheet as before with both feet. Tear the newspaper into two parts, and separate the two parts of the newspaper. Tear the first newspaper into small pieces with both feet. Remove the bunch of stubs and place them in a second, whole newspaper. Wrap everything into a ball shape with both feet. This step is enough to do once.

SUMMARY:
Subject will be trained to do regular foot exercise during their visit to the clinic. We will evaluate foot sensitivity and peripheral perfussion after

DETAILED DESCRIPTION:
Use an 8-10 MHz Doppler probe with a gel smeared over the sensor. Place the Doppler probe on the pulse area at a 45-60° angle to the skin surface.

Move the probe to find the most precise and robust arterial pulse before inflating the cuff.

The cuff is inflated about 20 mm Hg above the point where the arterial Doppler sound disappears.

Then slowly deflate until the Doppler sound reappears and records this value. The blood pressure at which the arterial pulse reappears is the systolic pressure for that blood vessel.

If the flow is still detected at the maximum inflation rate (300 mmHg), the cuff should be deflated immediately to avoid pain.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus Type 2

Exclusion Criteria:

* Chronic Heart Failure
* Chronic Kidney Diseae

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Fasting Blood Glucose | Cange Fasting Blood Glucose in 1 weeks
  Fasting Blood Glucose
Monofilament test | Cange monofilament test in 1 weeks
  Monofilament test to detect diabetic neuropathy
Ankle Brachial Index | Cange Ankle Brachial Index in 1 weeks
  Ankle Brachial Index

CONTACTS AND LOCATIONS:
Overall Officials: Nurhasan Agung Prabowo, MD, Principal Investigator — Universitas Sebelas Maret
Locations (1):
- RS UNS (Universitas Sebelas Maret Hospital), Surakarta, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No